CLINICAL TRIAL: NCT00010049
Title: Phase I/II Trial of STI571 (NSC 716051) in Patients With Recurrent Malignant Gliomas
Brief Title: Imatinib Mesylate in Treating Patients With Recurrent Malignant Glioma or Meningioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: NABTC-9908; CDR0000068437 (Registry Identifier: PDQ (Physician Data Query)); NCI-01-C-0243 (Other Grant/Funding Number: National Cancer Institute); UCLA-0101024; NCT00023179 (obsolete NCT alias)
Record Dates: First submitted 2001-02-02; First posted 2003-01-27 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult meningioma; adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult mixed glioma; adult pilocytic astrocytoma; adult subependymoma; adult grade III meningioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Meningioma; Glioblastoma; Astrocytoma; Oligodendroglioma; Glioma; Glioma, Subependymal; Gliosarcoma | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: imatinib mesylate

SUMMARY:
RATIONALE: Imatinib mesylate may interfere with the growth of tumor cells and may be an effective treatment for recurrent glioma and meningioma.

PURPOSE: Phase I/II trial to study the effectiveness of imatinib mesylate in treating patients who have progressive, recurrent, or unresectable malignant glioma or meningioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of imatinib mesylate in patients with recurrent malignant glioma or meningioma.
* Determine the safety profile of this drug in these patients.
* Determine the pharmacokinetics of this drug, with or without concurrent enzyme-inducing anti-epileptic drugs (EIAEDs), in these patients. (Stratum of patients currently taking EIAEDs closed to accrual as of 05/15/2003 for phase I and phase II)
* Determine angiogenic activity in vivo using functional neuro-imaging studies and in vitro with assays of serum angiogenic peptides.
* Determine the efficacy of this drug, in terms of 6-month progression-free survival and objective tumor response, in these patients.

OUTLINE: This is a multicenter, dose-escalation study. Patients are stratified according to concurrent enzyme-inducing anti-epileptic drug use (yes [stratum closed to accrual as of 05/15/2003 for phase I and phase II] vs no).

* Phase I (patients with glioma or meningioma) Patients in cohorts 1 and 2 receive oral imatinib mesylate (STI571) once daily on days 1-28. Patients in cohorts 3-5 receive oral STI571 twice daily on days 1 and 3-28 of the first course and on days 1-28 of subsequent courses. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of STI571 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II (patients with glioma) (glioblastoma multiforme patients excluded as of 05/15/2003) Patients receive oral STI571 at the MTD determined in phase I, 1-2 times daily for 4 weeks. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for phase I of the study within 6 months and a total of 39 patients will be accrued for phase II of the study within 6-8 months. (Glioblastoma multiforme patients excluded from phase II as of 05/13/2003).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed recurrent or unresectable malignant glioma

  * Glioblastoma multiforme (phase I only)
  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * Anaplastic mixed oligoastrocytoma
  * Malignant astrocytoma not otherwise specified
  * Gliosarcoma
  * Low-grade histology with subsequent diagnosis of malignant glioma allowed (phase I only) OR
* Histologically confirmed recurrent or unresectable benign or malignant meningioma (phase I only)
* No prior intracranial hemorrhage
* Failed prior radiotherapy
* Progressive or recurrent disease by MRI or CT scan and/or resection

  * PET or thallium scan, MR spectroscopy, or surgical documentation required in patients who have received prior interstitial brachytherapy or stereotactic radiosurgery
  * Stable dose of steroids for 5-7 days prior to MRI or CT scan

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* More than 8 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL (transfusion allowed)

Hepatic:

* Bilirubin less than 2 times upper limit of normal (ULN)
* SGOT less than 2 times ULN
* No significant hepatic disease

Renal:

* Creatinine less than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min
* No significant renal disease

Cardiovascular:

* No significant cardiac disease
* No deep venous or arterial thrombosis within the past 6 weeks

Pulmonary:

* No pulmonary embolism within the past 6 weeks

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for up to 6 months after study participation
* No other serious concurrent medical illness
* No serious active infection
* No concurrent disease that would obscure toxicity or alter drug metabolism
* No other malignancy within the past 3 years except nonmelanoma skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 1 week since prior interferon or thalidomide and recovered
* No concurrent immunotherapy
* No concurrent prophylactic filgrastim (G-CSF)

Chemotherapy:

* Recovered from prior chemotherapy
* At least 4 weeks since prior cytotoxic therapy
* At least 2 weeks since prior vincristine
* At least 6 weeks since prior nitrosoureas
* At least 4 weeks since prior temozolomide
* At least 3 weeks since prior procarbazine
* Prior polifeprosan 20 with carmustine implant (Gliadel wafer) allowed
* Prior radiosensitizers allowed
* No other concurrent chemotherapy
* Phase I only:

  * Prior chemotherapy required for anaplastic astrocytoma, anaplastic oligodendroglioma, and anaplastic mixed oligoastrocytoma
  * Prior treatment for up to 3 relapses allowed
* Phase II only:

  * Prior chemotherapy not required
  * Prior treatment for up to 2 relapses allowed

Endocrine therapy:

* See Disease Characteristics
* At least 1 week since prior tamoxifen and recovered
* No concurrent anticancer hormonal therapy

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* Recovered from prior surgical resection of recurrent or progressive disease

Other:

* At least 1 week since prior non-cytotoxic agents and recovered
* At least 1 week since prior tretinoin and recovered
* At least 2 weeks since prior drugs that affect hepatic metabolism
* No other concurrent investigational agents
* No concurrent warfarin

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2001-02-27 (Actual); Primary Completion 2005-03-17 (Actual); Study Completion 2006-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Y. Wen, MD, Study Chair — Dana-Farber Cancer Institute
Locations (11):
- United States (11):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- [Result] Wen PY, Yung WK, Lamborn KR, Dahia PL, Wang Y, Peng B, Abrey LE, Raizer J, Cloughesy TF, Fink K, Gilbert M, Chang S, Junck L, Schiff D, Lieberman F, Fine HA, Mehta M, Robins HI, DeAngelis LM, Groves MD, Puduvalli VK, Levin V, Conrad C, Maher EA, Aldape K, Hayes M, Letvak L, Egorin MJ, Capdeville R, Kaplan R, Murgo AJ, Stiles C, Prados MD. Phase I/II study of imatinib mesylate for recurrent malignant gliomas: North American Brain Tumor Consortium Study 99-08. Clin Cancer Res. 2006 Aug 15;12(16):4899-907. doi: 10.1158/1078-0432.CCR-06-0773. PMID 16914578
- [Result] Wen PY, Yung WKA, Lamborn K, et al.: Phase I/II study of imatinib mesylate (ST1571) for patients with recurrent malignant gliomas (NABTC 99-08). [Abstract] Neuro-Oncology 6 (4): TA-63, 385, 2004.